CLINICAL TRIAL: NCT00046423
Title: A Phase I Trial of ABI-007 Administered Weekly for Three Doses Every 4 Weeks in Patients With Advanced Non-hematologic Malignancies
Brief Title: A Trial of ABI-007 in Patients With Advanced Non-Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA-005-0
Record Dates: First submitted 2002-09-30; First posted 2002-10-03 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Neoplasms; Metastases, Neoplasm
Keywords: Cancer; solid tumor; Advanced malignancy; Taxane therapy; Biopsy-proven diagnosis of advanced malignancy; Various solid tumors which are refractory
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Albumin-Bound Paclitaxel

INTERVENTIONS:
Drug: ABI-007

SUMMARY:
This trial will treat patients with advanced (metastatic) cancer with a new chemotherapeutic agent that may be more readily tolerated than some standard therapies. Patients will be given the new chemotherapeutic medicine once a week, by intravenous route, for three weeks, followed by a rest week. Treatment will be repeated in four week cycles if the patient improves on the therapy, and if there are no adverse events that require withdrawal of medication.

DETAILED DESCRIPTION:
This will be a dose-escalating study. ABI-007 will be administered as an outpatient infusion for three weeks followed by a week of rest. The treatment course will repeat every 28 days. No pretreatment will normally be considered necessary. Patients will have white blood cell and platelet counts monitored as will indications of performance (Karnofsky Performance Status), and will be asked to describe adverse events, if present. Patients will be treated for a minimum of two cycles to be evaluable for the study, and may continue in the study for four cycles within the study, if tumor response and safety parameters warrant continuing. Patients may continue on study medication beyond this at the investigator's discretion.

ELIGIBILITY:
* At least 18 years of age
* Life expectancy of at least 2 months
* Off all therapy for at least 3 weeks prior to study drug administration
* Biopsy-proven diagnosis of advanced malignancy
* Patients with solid tumors who have failed standard therapy
* Karnofsky Performance Status of 70% or 0-2 SWOG Performance Status
* Hemoglobin at least 9
* White Blood Cell count of at least 3000/mm3 with absolute neutrophil count of at least 1500/mm3
* Platelet count of at least 100,000/mm3
* Serum Creatinine less than 2 mg/dL
* Transaminases less than 3X the upper limit of normal
* Patient must provide informed consent
* Serum Bilirubin less than 1.5 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2000-04

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Hawkins, M.D., Study Director — Celgene Corporation
Locations (1):
- Abraxis Bioscience, Inc., Durham, North Carolina, United States

REFERENCES:
- [Background] Nyman DW, Campbell KJ, Hersh E, Long K, Richardson K, Trieu V, Desai N, Hawkins MJ, Von Hoff DD. Phase I and pharmacokinetics trial of ABI-007, a novel nanoparticle formulation of paclitaxel in patients with advanced nonhematologic malignancies. J Clin Oncol. 2005 Nov 1;23(31):7785-93. doi: 10.1200/JCO.2004.00.6148. PMID 16258082